CLINICAL TRIAL: NCT02443324
Title: An Open-Label, Multicenter, Phase 1 Study of Ramucirumab Plus Pembrolizumab in Patients With Locally Advanced and Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma, Non-Small Cell Lung Cancer, Transitional Cell Carcinoma of the Urothelium, or Biliary Tract Cancer
Brief Title: A Study of Ramucirumab Plus Pembrolizumab in Participants With Gastric or GEJ Adenocarcinoma, NSCLC, Transitional Cell Carcinoma of the Urothelium, or Biliary Tract Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15787; I4T-MC-JVDF (Other: Eli Lilly and Company); 2015-001473-40 (EudraCT Number); KEYNOTE -098 (Other: Merck)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Gastric Adenocarcinoma; Adenocarcinoma of the Gastroesophageal Junction; Non-small Cell Lung Cancer; Carcinoma, Transitional Cell; Biliary Tract Cancer
Keywords: immuno-oncology; Vascular Endothelial Growth Factor (VEGF); angiogenesis; PD-1; carcinoma of the bladder; carcinoma of the urethra; carcinoma of the ureter; carcinoma of the renal pelvis; carcinoma of the biliary tract
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Biliary Tract Neoplasms; Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms | interventions — Ramucirumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Cohort A (Experimental): Participants with gastroesophageal junction (GEJ) cancer [Second-Third Line (L)] received 8 milligrams per kilogram (mg/kg) ramucirumab given intravenously (IV) on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 for every 3 weeks (Q3W) of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Cohort A1 (Experimental): Participants with BTC cancer (Second-Third L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab
- Cohort A2 (Experimental): Participants with Gastric-GEJ cancer (First L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Cohort B (Experimental): Participants with Gastric-GEJ cancer (Second-Third L) received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Cohort C (Experimental): Participants with NSCLC (Second-Fourth L) received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Cohort D (Experimental): Participants with Urothelial cancer (Second-Fourth L) received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab
- Cohort E (Experimental): Participants with NSCLC cancer (First L) received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza
Drug: Pembrolizumab — Administered IV
  Other Names: MK3475
  Arms: Cohort A; Cohort A2; Cohort B; Cohort C; Cohort D; Cohort E

SUMMARY:
The main purpose of this study is to evaluate the safety and preliminary efficacy of the combination of the study drug known as ramucirumab plus pembrolizumab in participants with locally advanced and unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma, non-small cell lung cancer (NSCLC), transitional cell carcinoma of the urothelium, or biliary tract cancer (BTC).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease or locally advanced, unresectable disease.

  * Has histopathologically confirmed gastric or GEJ adenocarcinoma with documented disease progression after 0-2 prior lines of systemic therapy
  * Has histopathologically confirmed nonsquamous or squamous NSCLC with documented disease progression after 0-3 prior lines of systemic therapy
  * Has histopathologically confirmed transitional cell carcinoma of the urothelium (bladder, urethra, or renal pelvis) with documented disease progression after 1-3 prior lines of systemic therapy
  * Has histologically confirmed biliary tract adenocarcinoma with documented progression after 1-2 prior lines of systemic therapy
* Availability of tumor tissue for biomarker analysis from a newly obtained core or excisional biopsy or willing to undergo a tumor biopsy. For first line NSCLC participants only, PD-L1 expression should be 1% or higher.
* Have an Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Has adequate organ function.
* Have an anticipated life expectancy of ≥3 months.

Exclusion Criteria:

* Have known brain metastases.
* Has received ≥3 lines of prior systemic therapy for gastric or GEJ adenocarcinoma and BTC or ≥4 lines for NSCLC or urothelial cancer.
* Has active autoimmune disease.
* Known human immunodeficiency virus (HIV) infection.
* Known active hepatitis B or hepatitis C infection.
* Has received any previous systemic therapy targeting vascular endothelial growth factor (VEGF) or VEGF receptor, or programmed death (PD) 1 or PD-ligand 1/2 signaling pathways.
* Have received a live vaccine within 30 days prior to enrollment. Seasonal flu vaccines that do not contain live virus are permitted.
* Have had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Have an elective or a planned major surgery during the course of the trial or has undergone major surgery within 28 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- United States (7):
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Japan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamanashi
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manchester
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sutton

REFERENCES:
- [Derived] Herbst RS, Arkenau HT, Bendell J, Arrowsmith E, Wermke M, Soriano A, Penel N, Santana-Davila R, Bischoff H, Chau I, Mi G, Wang H, Rasmussen E, Ferry D, Chao BH, Paz-Ares L. Phase 1 Expansion Cohort of Ramucirumab Plus Pembrolizumab in Advanced Treatment-Naive NSCLC. J Thorac Oncol. 2021 Feb;16(2):289-298. doi: 10.1016/j.jtho.2020.10.004. Epub 2020 Oct 15. PMID 33068794
- [Derived] Herbst RS, Arkenau HT, Santana-Davila R, Calvo E, Paz-Ares L, Cassier PA, Bendell J, Penel N, Krebs MG, Martin-Liberal J, Isambert N, Soriano A, Wermke M, Cultrera J, Gao L, Widau RC, Mi G, Jin J, Ferry D, Fuchs CS, Petrylak DP, Chau I. Ramucirumab plus pembrolizumab in patients with previously treated advanced non-small-cell lung cancer, gastro-oesophageal cancer, or urothelial carcinomas (JVDF): a multicohort, non-randomised, open-label, phase 1a/b trial. Lancet Oncol. 2019 Aug;20(8):1109-1123. doi: 10.1016/S1470-2045(19)30458-9. Epub 2019 Jul 10. PMID 31301962
- [Derived] Arkenau HT, Martin-Liberal J, Calvo E, Penel N, Krebs MG, Herbst RS, Walgren RA, Widau RC, Mi G, Jin J, Ferry D, Chau I. Ramucirumab Plus Pembrolizumab in Patients with Previously Treated Advanced or Metastatic Biliary Tract Cancer: Nonrandomized, Open-Label, Phase I Trial (JVDF). Oncologist. 2018 Dec;23(12):1407-e136. doi: 10.1634/theoncologist.2018-0044. Epub 2018 May 31. PMID 29853658
- See also: A Study of Ramucirumab Plus Pembrolizumab in Participants With Gastric or GEJ Adenocarcinoma, NSCLC, Transitional Cell Carcinoma of the Urothelium, or Biliary Tract Cancer — https://trials.lilly.com/en-US/trial/98852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study has Phase 1a (dose-limiting toxicity [DLT] observation) and expansion Phase 1b (safety and preliminary efficacy) included participants with 2 dosing schedules:
  Schedule 1: gastroesophageal junction (GEJ) cancer (Cohorts A, A2) and biliary tract cancer (Cohorts A1); Schedule 2: Gastric-GEJ cancer (Cohort B), nonsmall cell lung cancer (NSCLC) (Cohorts C, E), and urothelial cancer (Cohort D).
Pre-assignment Details: Participants who did not "complete" study were those who discontinued study treatment by the time of study completion.
Groups:
- Cohort A: Participants with Gastric-GEJ cancer [Second-Third Line (L)] received 8 milligrams per kilogram (mg/kg) ramucirumab given intravenously (IV) on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 for every 3 weeks (Q3W) of a 21-day cycle.
Period: Overall Study
Arm/Group | Cohort A | Cohort A1 | Cohort A2 | Cohort B | Cohort C | Cohort D | Cohort E
Started | 24 | 26 | 29 | 17 | 28 | 24 | 27
Received at Least One Dose of Study Drug | 24 | 26 | 28 | 17 | 27 | 24 | 26
Phase 1a | 8 | 0 | 0 | 0 | 3 | 0 | 0
Phase 1b | 16 | 26 | 28 | 17 | 24 | 24 | 26
Completed | 0 | 1 | 4 | 1 | 7 | 0 | 8
Not Completed | 24 | 25 | 25 | 16 | 21 | 24 | 19
Not completed — Death | 4 | 1 | 0 | 3 | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 3 | 5 | 1 | 1 | 0 | 2
Not completed — Progressive Disease | 20 | 20 | 13 | 10 | 13 | 17 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 3 | 0 | 4 | 3 | 3
Not completed — Enrolled but Never Treated | 0 | 0 | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Cohort A: Participants with Gastric-GEJ cancer (Second-Third L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort A1 | Cohort A2 | Cohort B | Cohort C | Cohort D | Cohort E | Total
Number analyzed (Participants) | 24 | 26 | 28 | 17 | 27 | 24 | 26 | 172
Age, Continuous [Mean (Full Range); unit: years] | 56.0 [24.0 to 78.0] | 62.5 [36.0 to 78.0] | 63.0 [31.0 to 83.0] | 61.0 [28.0 to 73.0] | 65.0 [34.0 to 82.0] | 63.0 [45.0 to 87.0] | 63.0 [42.0 to 85.0] | 61.28 [24.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 7 | 3 | 6 | 10 | 14 | 65
  Male | 17 | 8 | 21 | 14 | 21 | 14 | 12 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 3 | 2 | 3 | 4 | 0 | 20
  Not Hispanic or Latino | 20 | 19 | 16 | 12 | 21 | 10 | 25 | 123
  Unknown or Not Reported | 2 | 1 | 9 | 3 | 3 | 10 | 1 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 4
  White | 19 | 23 | 17 | 16 | 26 | 22 | 22 | 145
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 10 | 0 | 0 | 2 | 3 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 11 | 8 | 4 | 8 | 11 | 47
  United Kingdom | 15 | 11 | 7 | 5 | 2 | 5 | 6 | 51
  France | 2 | 3 | 7 | 1 | 8 | 2 | 2 | 25
  Germany | 0 | 1 | 1 | 0 | 0 | 1 | 5 | 8
  Spain | 4 | 9 | 2 | 3 | 13 | 8 | 2 | 41

OUTCOME MEASURES:

1. Primary Outcome: Phase 1a: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: DLT is defined as an Adverse Event (AE) that is likely related to study medication or combination,and fulfills any one of following criteria:Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0): Grade (Gr) 3 and 4 nonlaboratory toxicity (tox),Any Gr 3 or 4 laboratory value if medical intervention is required to treat participant (pt) or abnormality persists for >1 week;Hematologic tox:Gr 4 toxicity lasting ≥ 7 days,or Gr 3 thrombocytopenia if associated with bleeding and requires platelet transfusion,or Febrile neutropenia Gr 3 or Gr 4;GR 5 tox (death);Any toxicity that is possibly related to study treatment that requires withdrawal of pt from study during Cycle 1,A delay of > 14 days due to persistent Grade ≥ 2 toxicities in initiating Cycle 2,with exception of Grade 2 fatigue;Any infusion or hypersensitivity reactions are NOT a DLT. A summary of other nonserious AEs and all Serious AEs,regardless of causality is located in Reported Adverse Event section.
Time Frame: Cycle 1 (21 Days)
Population: All enrolled participants who received at least one dose of the study drug in dose escalation phase and experienced a DLT. DLT was assessed in Phase 1a of Cohorts A and C during Cycle 1.
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort C
Number analyzed (Participants) | 6 | 3
participants | 1 | 0

2. Secondary Outcome: Phase 1a and 1b: Percentage of Participants Who Achieve Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants per cohort with at least 1 measurable lesion, multiplied by 100. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease (Up to 24 Months)
Population: All enrolled participants who received at least one dose of the study drug. Per Protocol, Cohort A and B participants [Gastric-GEJ cancer (Second-Third L)] were combined and outcome data was analyzed under a single arm (Cohort A and B).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A and B: Participants with Gastric-GEJ cancer (Second-Third L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle in Cohort A.
  Participants with Gastric-GEJ cancer (Second-Third L) received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle in Cohort B.
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 41 | 26 | 28 | 27 | 24 | 26
percentage of participants | 7.3 [1.5 to 19.9] | 3.8 [0.1 to 19.6] | 25.0 [10.7 to 44.9] | 29.6 [13.8 to 50.2] | 12.5 [2.7 to 32.4] | 42.3 [23.4 to 63.1]

3. Secondary Outcome: Phase 1a and 1b: Percentage of Participants Who Exhibit Stable Disease (SD) or CR or PR [Disease Control Rate (DCR)]
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. Participants who do not have any postbaseline tumor response assessments for any reason were considered.
Time Frame: Baseline to Measured Progressive Disease (Up to 24 Months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 41 | 26 | 28 | 27 | 24 | 26
percentage of participants | 51.2 [35.1 to 67.1] | 38.5 [20.2 to 59.4] | 67.9 [47.6 to 84.1] | 85.2 [66.3 to 95.8] | 50.0 [29.1 to 70.9] | 84.6 [65.1 to 95.6]

4. Secondary Outcome: Phase 1a and 1b: Duration of Response (DoR)
Description: The duration of response is defined only for responders (patients with a confirmed CR or PR). It is measured from the date of first evidence of a confirmed CR or PR to the date of objective progression or the date of death due to any cause, whichever is earlier. If a responder is not known to have died or have objective progression as of the data inclusion cutoff date, DoR will be censored at the date of the last complete objective progression-free disease assessment (CR or PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Up to 24 Months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 3 | 1 | 7 | 8 | 3 | 11
months | 6.7 [4.4 to 17.5] | 6.0 [NA to NA] — Only 1 participant had PR, therefore 95% Confidence Interval was not calculable. | NA [9.7 to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate. | NA [11.1 to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate. | 8.3 [4.6 to 16.8] | NA [5.2 to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate.

5. Secondary Outcome: Phase 1a and 1b: Time to First Response (TTR)
Description: TTR is defined as the time from the date of first study treatment until the first evidence of a confirmed CR or PR.
Time Frame: Baseline to Date of CR or PR (Up to 24 Months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 3 | 1 | 7 | 8 | 3 | 11
months | 1.4 [1.4 to 4.1] | 2.7 [NA to NA] — Only 1 participant had PR, therefore 95% Confidence Interval was not calculable. | 2.7 [1.3 to 2.8] | 2.1 [1.3 to 3.0] | 2.8 [1.3 to 5.5] | 1.4 [1.2 to 3.0]

6. Secondary Outcome: Phase 1a and 1b: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first study treatment until the date of the first observed radiographically documented progressive disease (PD) or death due to any cause, whichever is earlier. PD was determined using RECIST criteria. PD is ≥20% increase in sum of longest diameter of target lesions and/or a new lesion.
Time Frame: Baseline to PD or Death of Any Cause (Up to 24 Months)
Population: All enrolled participants who received at least one dose of the study drug. Censored participants: Cohort A and B = 3; Cohort A1 = 4; Cohort A2 = 8; Cohort C = 10; Cohort D = 3 and Cohort E = 13. Per Protocol, Cohort A and B participants [Gastric-GEJ cancer (Second-Third L)] were combined and outcome data was analyzed under a single arm (Cohort A and B).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 41 | 26 | 28 | 27 | 24 | 26
months | 2.5 [1.5 to 4.2] | 1.6 [1.4 to 2.8] | 5.6 [2.7 to 11.5] | 9.7 [4.6 to 27.6] | 1.9 [1.2 to 2.8] | 9.3 [4.0 to NA] — upper 95% confidence interval was not achieved due to high censoring rate.

7. Secondary Outcome: Phase 1a and 1b: Overall Survival (OS)
Description: The OS time is defined as the time from baseline to the date of death from any cause. If a participant is not known to have died on or before the date of data cut-off, OS data will be censored on the last date (on or before the cut-off date) the participant was known to be alive.
Time Frame: Baseline to Death from Any Cause (Up to 24 Months)
Population: All enrolled participants who received at least one dose of the study drug. Censored participants: Cohort A and B = 8; Cohort A1 = 8; Cohort A2 = 12; Cohort C = 12; Cohort D = 6 and Cohort E = 18. Per Protocol, Cohort A and B participants [Gastric-GEJ cancer (Second-Third L)] were combined and outcome data was analyzed under a single arm (Cohort A and B).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A and B | Cohort A1 | Cohort A2 | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 41 | 26 | 28 | 27 | 24 | 26
months | 5.9 [4.4 to 10.6] | 6.4 [4.2 to 13.3] | 14.6 [5.4 to NA] — upper 95% confidence interval was not achieved due to high censoring rate. | 26.2 [11.8 to NA] — upper 95% confidence interval was not achieved due to high censoring rate. | 6.4 [2.5 to 18.7] | NA [13.2 to NA] — Median and the upper 95% confidence interval was not achieved due to high censoring rate.

8. Secondary Outcome: Phase 1a and 1b: Pharmacokinetics (PK): Minimum Trough Concentration (Cmin) of Ramucirumab
Description: PK: Cmin of Ramucirumab following administration every 3 weeks.
Time Frame: Phase 1a (Gastric-GEJ or BTC participants (pts)): Week (Wk) 1, 3, 6 and 9; Phase 1a (Gastric, NSCLC, or urothelial pts): Wk 3, 6, 9 and 12; Cohort A, A1, A2: Wk 1, 3, 6, 9, 12, 18, 19 and 24; Cohort B,C,D,E: Wk 3, 6, 9, 12, 18, 19 and 24
Population: All enrolled participants who received at least one dose of the study drug and had evaluable ramucirumab PK data. PK was assessed both in Phase 1a and 1b as per protocol analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (μg/mL)
Groups:
- Phase 1a: Gastric-GEJ or BTC: Participants received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
- Phase 1 a: Gastric, NSCLC, or Urothelial Patients: Participants received 10 mg/kg ramucirumab given IV on day 1 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
- Cohort B: Participants with Gastric-GEJ cancer (Second-Third L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
Arm/Group | Phase 1a: Gastric-GEJ or BTC | Phase 1 a: Gastric, NSCLC, or Urothelial Patients | Cohort A | Cohort A1 | Cohort A2 | Cohort B | Cohort C | Cohort D | Cohort E
Number analyzed (Participants) | 6 | 3 | 16 | 22 | 26 | 15 | 23 | 15 | 21
micrograms/milliliter (μg/mL)
  Week 1: number analyzed (Participants) | 6 | 0 | 16 | 22 | 26 | 0 | 0 | 0 | 0
  Week 1 | 50.9 (24) |  | 44.2 (28) | 45.2 (41) | 45.9 (23) |  |  |  |
  Week 3: number analyzed (Participants) | 5 | 3 | 11 | 20 | 22 | 15 | 23 | 15 | 21
  Week 3 | 52 (29) | 20.9 (35) | 40 (48) | 44.1 (57) | 45.2 (32) | 13.3 (93) | 22.5 (62) | 20.9 (54) | 15.6 (70)
  Week 6: number analyzed (Participants) | 5 | 2 | 5 | 11 | 18 | 12 | 15 | 15 | 18
  Week 6 | 69 (29) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 21.2 μg/mL, 30.6 μg/mL | 79.8 (30) | 69.1 (68) | 61 (38) | 25.7 (74) | 33.8 (68) | 23.3 (102) | 19.3 (115)
  Week 9: number analyzed (Participants) | 2 | 3 | 8 | 6 | 13 | 9 | 18 | 11 | 15
  Week 9 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 45.6 μg/mL, 72.5 μg/mL | 32.7 (20.6) | 72.8 (46) | 94.3 (40) | 78.8 (31) | 32.7 (60) | 40.1 (63) | 34.8 (73) | 28.6 (90)
  Week 12: number analyzed (Participants) | 0 | 2 | 5 | 2 | 10 | 8 | 16 | 8 | 10
  Week 12 |  | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 26.9 μg/mL, 38.7 μg/mL | 89.3 (35) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 140 μg/mL, 160 μg/mL | 80.2 (38) | 36.8 (48) | 47.1 (45) | 34.9 (141) | 26.3 (89)
  Week 18: number analyzed (Participants) | 0 | 0 | 5 | 2 | 7 | 4 | 11 | 5 | 9
  Week 18 |  |  | 92.4 (71) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 147 μg/mL, 171 μg/mL | 87.6 (48) | 52.7 (45) | 44.4 (31) | 52.6 (36) | 37.1 (66)
  Week 19: number analyzed (Participants) | 0 | 0 | 3 | 1 | 5 | 0 | 0 | 0 | 0
  Week 19 |  |  | 149 (69) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =1. Individual value = 215 μg/mL | 120 (34) |  |  |  |
  Week 24: number analyzed (Participants) | 0 | 0 | 3 | 1 | 3 | 4 | 10 | 2 | 7
  Week 24 |  |  | 116 (83) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =1. Individual value = 178 μg/mL | 95.7 (27) | 43.6 (40) | 45 (29) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as n =2. Individual values = 39.5 μg/mL, 88 μg/mL | 42.1 (87)

ADVERSE EVENTS:
Time Frame: Baseline Up to 5.9 Years
Description: All enrolled participants who received at least one dose of the study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Cohort C: Participants with NSCLC (Second-Fourth L) received 8 mg/kg ramucirumab given IV on day 1 and 8 in combination with 200 mg pembrolizumab given IV on day 1 Q3W of a 21-day cycle.
Arm/Group | Cohort A | Cohort A1 | Cohort A2 | Cohort B | Cohort C | Cohort D | Cohort E
All-Cause Mortality (participants affected / at risk) | 21/24 | 19/26 | 17/28 | 13/17 | 16/27 | 18/24 | 9/26
Serious Adverse Events (participants affected / at risk) | 10/24 | 15/26 | 16/28 | 10/17 | 15/27 | 16/24 | 14/26
Other Adverse Events (participants affected / at risk) | 23/24 | 26/26 | 28/28 | 16/17 | 27/27 | 24/24 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=24) | Cohort A1 (N=26) | Cohort A2 (N=28) | Cohort B (N=17) | Cohort C (N=27) | Cohort D (N=24) | Cohort E (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraneoplastic encephalomyelitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A (N=24) | Cohort A1 (N=26) | Cohort A2 (N=28) | Cohort B (N=17) | Cohort C (N=27) | Cohort D (N=24) | Cohort E (N=26)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (4) | 5 (16) | 3 (15) | 5 (5) | 2 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (3) | 0 (0) | 1 (3) | 2 (4) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 8 (11) | 2 (2) | 2 (3)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 9 (11) | 5 (7) | 4 (4) | 3 (4) | 4 (5) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (3) | 5 (6) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 5 (7) | 2 (6) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (7) | 5 (6) | 5 (6) | 8 (10) | 4 (4) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 9 (13) | 11 (28) | 6 (8) | 8 (20) | 7 (11) | 8 (9)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 6 (10) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (9) | 11 (12) | 12 (14) | 2 (2) | 5 (11) | 5 (6) | 8 (11)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (5) | 5 (6) | 5 (6) | 1 (1) | 4 (11) | 0 (0) | 2 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 5 (5) | 7 (12) | 2 (5) | 4 (8) | 4 (5) | 3 (3)
Asthenia (General disorders) | 1 (5) | 4 (9) | 2 (6) | 2 (7) | 8 (31) | 0 (0) | 4 (5)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 14 (21) | 9 (12) | 19 (33) | 9 (15) | 10 (11) | 11 (12) | 9 (15)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 3 (4) | 2 (2) | 8 (14) | 4 (6) | 4 (16) | 3 (3) | 5 (6)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 3 (4) | 1 (2)
Pyrexia (General disorders) | 2 (2) | 6 (7) | 0 (0) | 3 (5) | 4 (4) | 6 (6) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4) | 3 (3) | 2 (3) | 2 (3) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 3 (7) | 1 (1) | 3 (3) | 5 (6) | 6 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (7) | 3 (3) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (18) | 5 (11) | 0 (0) | 4 (6) | 4 (5) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (14) | 6 (12) | 1 (2) | 5 (6) | 4 (5) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (6) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 0 (0)
Mammogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 3 (6) | 5 (7) | 4 (5) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (11) | 7 (9) | 9 (15) | 4 (4) | 10 (15) | 8 (10) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (4) | 0 (0) | 2 (4) | 0 (0) | 1 (3)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (7) | 3 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (22) | 1 (3) | 2 (3) | 2 (6) | 2 (8) | 1 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tetany (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 3 (4) | 0 (0) | 9 (19) | 2 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 3 (7) | 1 (1) | 6 (8) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (5) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 4 (5) | 3 (4) | 1 (1) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (6) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 5 (6) | 8 (13) | 2 (3) | 5 (9) | 5 (6) | 4 (5)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 5 (6) | 8 (28) | 0 (0) | 4 (15) | 5 (10) | 4 (9)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0/7 (0) | 1/18 (1) | 0/7 (0) | 1/3 (1) | 0/6 (0) | 0/10 (0) | 0/14 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1/17 (1) | 0/8 (0) | 0/21 (0) | 0/14 (0) | 0/21 (0) | 0/14 (0) | 0/12 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0/7 (0) | 1/18 (1) | 0/7 (0) | 0/3 (0) | 0/6 (0) | 0/10 (0) | 1/14 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 4 (4) | 3 (3) | 11 (21) | 2 (2) | 6 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2) | 8 (11) | 3 (3) | 8 (11) | 1 (1) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 6 (7) | 2 (2) | 5 (7) | 1 (1) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 3 (4) | 0 (0) | 0 (0) | 4 (8) | 2 (2) | 6 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 2 (3) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 3 (8) | 2 (2) | 0 (0) | 0 (0) | 5 (11)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (10) | 9 (26) | 10 (22) | 4 (8) | 9 (12) | 7 (9) | 6 (15)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT02443324/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02443324/SAP_001.pdf